CLINICAL TRIAL: NCT06326801
Title: Effect of Resistive Diaphragmatic Breathing Exercise With Pursed Lips Breathing Exercise on Pulmonary Function, Trunk Control and Functional Capacity in Sub-acute Stroke Patients
Brief Title: Resistive Diaphragmatic Breathing Exercise With Pursed Lips Breathing Exercise in Sub-acute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/014220 Muhammad Iqbal
Record Dates: First submitted 2024-01-18; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A (Active Comparator): 1. Resistive Diaphragmatic breathing exercise
  2. Pursed lips breathing exercise
  3. Conventional stroke physiotherapy
  Interventions: Other: Resistive Diaphragmatic breathing exercise; Other: Diaphragmatic breathing exercise; Other: Conventional stroke physiotherapy
- Treatment B (Active Comparator): 1. Diaphragmatic breathing exercise
  2. Pursed lips breathing exercise
  3. Conventional stroke physiotherapy
  Interventions: Other: Resistive Diaphragmatic breathing exercise; Other: Diaphragmatic breathing exercise; Other: Conventional stroke physiotherapy
- Control group (Active Comparator): a) Conventional stroke physiotherapy
  Interventions: Other: Resistive Diaphragmatic breathing exercise; Other: Diaphragmatic breathing exercise; Other: Conventional stroke physiotherapy

INTERVENTIONS:
Other: Resistive Diaphragmatic breathing exercise — 1. Resistive Diaphragmatic breathing exercise
  2. Pursed lips breathing exercise
  3. Conventional stroke physiotherapy
Other: Diaphragmatic breathing exercise — 1. Diaphragmatic breathing exercise
  2. Pursed lips breathing exercise
  3. Conventional stroke physiotherapy
Other: Conventional stroke physiotherapy — Conventional stroke physiotherapy

SUMMARY:
To determine whether resistive diaphragmatic breathing exercise with pursed lips breathing exercise improve pulmonary function in sub-acute ischemic stroke, To determine whether resistive diaphragmatic breathing exercise with pursed lips breathing exercise improve Trunk Control in sub-acute ischemic stroke, To determine whether resistive diaphragmatic breathing exercise with pursed lips breathing exercise improve Functional Capacity in sub-acute ischemic stroke

ELIGIBILITY:
Inclusion Criteria

* Age 40-65 years
* Onset of ischemic stroke in first two week
* First episode of unilateral stroke with hemiparesis during previous 12 months
* Patient with no serious cognitive deficits i-e mini-mental state examination (score >22) ability to understand, perform and follow simple verbal instructions
* Functional ambulation category (FAC) >3
* 6 min walk test distance should be >200 m

Exclusion Criteria:

* Known case of cardiopulmonary disease, BP > 180/100 mmHg twice in 24 hours
* Known case of neurological disease other than stroke, Known case of orthopedic disease i-e funnel chest, rib fractures or any other orthopedic deformity
* Medication that would influence metabolic or cardiorespiratory responses to exercise Impaired level of consciousness, Evidence of gross cognitive impairment.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
pulmonary function | 4 weeks
  The pulmonary functions Spirometer measure can be expressed as Forced Expiratory Volume in 1 second (FEV1) and Force Vital Capacity (FVC) .
Trunk Control | 4weeks
  Trunk performance and coordination by static and dynamic sitting balance was measured by TIS.TIS comprises 17 items, measures dynamic and static sitting balance and trunk co-ordination. The TIS total score is 0-23 points, higher scores show better performance.
  It takes about 6 to 16 minutes in applying TIS
Functional Capacity | 4weeks
  6 MWT is used for functional capacity of participants, by walking for 6 minutes.
  Participant walk between the point marked, as numerous periods as can in 6 minutes.
  The 6-minute walk (6mw) test is a reliable and valid measure of for assessing functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Razzaq, MS, Principal Investigator — Riphah International University
Locations (1):
- Northwest General Hospital, Peshawar;, Peshawar, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No